CLINICAL TRIAL: NCT06507761
Title: Comparison of the Short-term Effect of Superficial Thermotherapy Applications in Acute Nonspecific Neck Pain-Randomised Controlled Trial
Brief Title: Thermotherapy in Acute Nonspecific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc, Prof. Nuray Alaca, Head of department Physiotherapy and Rehabilitation, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/9/340
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Cold
MeSH Terms: conditions — Neck Pain; Common Cold | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Group (Sham Comparator)
  Interventions: Other: Sham
- Hot Pack Group (Active Comparator)
  Interventions: Other: Hot Pack
- Cold Pack Group (Active Comparator)
  Interventions: Other: Cold Pack

INTERVENTIONS:
Other: Sham — An unrefrigerated room temperature Cold Pack will be wrapped in a towel and applied to the patient's posterior neck and back for 15 minutes while the patient is lying face down.
  Arms: Sham Group
Other: Hot Pack — Hot pack (55-60 degrees) application will be wrapped in a towel and applied to the back side neck and back of the patient for 15 minutes while the patient is lying face down.
  Arms: Hot Pack Group
Other: Cold Pack — Cold pack application (2-4 degrees) will be wrapped in a towel and applied to the patient's back side neck and back for 15 minutes while the patient is lying prone.
  Arms: Cold Pack Group

SUMMARY:
Neck pain is one of the most common musculoskeletal pain disorders secondary to low back pain. Medical and non-medical treatments such as physiotherapy are applied in its treatment. Patients with nonspecific neck pain (NBA) can be treated with various interventions such as drug therapy, manual therapy, heat and exercise. Although it is frequently used in clinical practice, there is no evidence that superficial thermotherapy (hot or cold) methods effectively relieve neck pain. Therefore, this study aims to compare the short-term effects of superficial hot or cold applications on pain, range of motion and functional status in patients with NBA.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with nonspecific neck pain by a doctor,
* To be between the ages of 18-65,
* Neck pain lasting for less than 1 month
* No previous neck or shoulder surgery,
* No shoulder pain due to any cause,
* A tumour or inflammatory disease underlying the neck pain not to be found,
* A clinically underlying stenosis or discogenic problem not to be present.
* Negative results from the following clinical examination tests;

Spurling test, Lhermitte test, Cervical distraction test, Adson test,

Exclusion Criteria:

* Not meeting the inclusion criteria,
* Positive neurological examination (positive motor presence, reflex or sensory abnormalities indicating spinal root compression) or abnormal neurological findings related to nerve compression in the upper limb
* Systemic rheumatological or metabolic diseases or cancer
* Refusal to participate in the study,
* Failure to complete treatment,
* Having any neurological problem
* Severe psychological illnesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NPRS-11) | Change from baseline pain score at 3th day
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
Range of Motion | Change from baseline range of motion at 3th day
  CROM device will be used. The active range of motion of each individual will be measured and measured in accordance with the manufacturer's procedures
Global Rating of Change scale (Patient Satisfaction) | Change from baseline Global Rating of Change scale at 3th day
  Patient satisfaction regarding improvement in shoulder function will be evaluated by the Global Rating of Change scale. All participants will be asked to rate their condition after a six-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly between -3 to +3, with a higher value indicating better condition in this study.

SECONDARY OUTCOMES:
Neck disability index | Change from baseline disability scale at 3th day
  Since some parts of the 10-item questionnaire could not be answered by the patients (driving, working life), the average neck disability index score will be calculated by dividing the total score by the number of questions answered. The scoring is between 0 and 50. 0 points means the best result, 50 points means the worst result. 0 - 4 points; no disability, 5 - 14 points; mild disability, 15 - 24 points; moderate disability, 25 - 34 points; severe disability, > 35 points; complete disability
Pressure Pain Threshold | Change from baseline Pressure Pain Threshold at 3th day
  A digital pressure algometer will be applied to the web space of the foot opposite the trigger point. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Nuray ALACA, Istanbul
  - Acibadem University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided